CLINICAL TRIAL: NCT06048601
Title: A Multi-center Phase 3 Study of 18F-florbetaben Positron Emission Tomography/Computed Tomography (PET-CT) to Non-invasively Diagnose Cardiac AL Amyloidosis
Brief Title: 18F-florbetaben PET-CT to Non-invasively Diagnose Cardiac AL Amyloidosis
Acronym: PETAL
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Toscana Gabriele Monasterio (Other)
Responsible Party: Principal Investigator, Michele Emdin, MD, PhD, FESC, FHFA, Fondazione Toscana Gabriele Monasterio
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PETAL2023
Record Dates: First submitted 2023-09-16; First posted 2023-09-21 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Amyloid; Amyloid Cardiomyopathy
MeSH Terms: conditions — Alzheimer Disease; Amyloid Neuropathies, Familial

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- two diagnostic approaches to the diagnosis of AL-CA in patients with a monoclonal protein (Experimental): traditional invasive approach vs. non-invasive approach using the visual assessment of 18F-florbetaben PET/TC
  Interventions: Diagnostic Test: 18F-florbetaben PET/CT

INTERVENTIONS:
Diagnostic Test: 18F-florbetaben PET/CT — 18F-florbetaben positron emission tomography/computed tomography

SUMMARY:
Amyloidoses are systemic or acquired disorders characterized by the deposition in the extracellular spaces of amyloid fibers formed by proteins codified by mutated genes or non-mutated but misfolded proteins. Cardiac involvement in amyloidosis is an important determinant of the clinical presentation and can be found in patients with amyloid light-chain (AL) or transthyretin (ATTR) amyloidosis, the latter due to the deposition of normal proteins (formerly known as senile amyloidosis) or mutated proteins. Cardiac amyloidosis (CA) has a poor prognosis that further worsens if the diagnosis and treatment are delayed. Nuclear medicine techniques have emerged as important tools for the diagnosis and characterization of CA. It has been recently demonstrated that cardiac uptake of bone tracers allows to identify the deposition of transthyretin in the heart, while it is not useful for the diagnosis of AL-CA, which currently requires the histological demonstration of amyloid fibers in a tissue sample taken with invasive procedures such as an endomyocardial biopsy. Recently, some PET tracers developed to identify beta-amyloid deposits in the brain proved able to detect an uptake even in the heart; nonetheless their possible use to diagnose CA is still debated. One of those tracers is florbetaben labelled with 18F, which displays a high binding affinity with beta-amyloid in the brain, while the experience on its use to identify extracranial amyloid deposits is still limited. Three studies have reported a cardiac uptake of 18F-florbetaben in AL or ATTR amyloidosis. Tracer uptake could be detected starting from 15 minutes after tracer administration. In a case series of 60 patients (20 with AL-CA, 20 with ATTR-CA and 20 with CA suspected but excluded) we demonstrated that the evidence of a myocardial uptake in a late acquisition can effectively discriminate AL- from ATTR-CA or other conditions. Indeed, patients with AL-CA displayed an intense and persistent myocardial uptake in static acquisitions at all time points, while patients with ATTR-CA and those without CA displayed a rapid reduction of the uptake after the early acquisition.

This study aims to compare the performance of PET/CT with 18F-florbetaben to diagnose AL-CA compared with the current diagnostic standard, which requires a tissue biopsy.

Primary objective:

To define the agreement (with its 95% confidence interval) between two diagnostic approaches to the diagnosis of AL-CA in patients with a monoclonal protein: the traditional invasive approach and a non-invasive approach using the visual assessment of 18F-florbetaben PET/TC.

Secondary objectives:

* To define the diagnostic performance of PET/CT with 18F-florbetaben (visual evaluation) in terms of sensitivity, specificity, positive and negative predictive value;
* To define cut-offs from myocardial uptake quantification to confirm or discard AL-CA among patients with suspected CA and a monoclonal protein, compared to the standard diagnostic algorithm, from quantitative uptake values;
* To assess the changes in the degree of myocardial 18F-florbetaben uptake over 12 months in patients with AL-CA;
* To assess the safety and tolerability of PET/CT with 18F-florbetaben in patients evaluated for suspected CA.

ELIGIBILITY:
Inclusion Criteria:

* Men and women aged >18 years;
* Ability to understand, sign and date the informed consent;
* NT-proBNP values> 332 ng/L in the absence of renal in-sufficiency or atrial fibrillation or mean left ventricular wall thickness >12 mm on echocardiogram and / or a pat-tern of circumferential or diffuse late gadolinium en-hancement and/or BNP >81 ng/L, in a clinical setting seemed compatible with CA by experienced doctors.

Exclusion Criteria:

* Hypersensitivity to the active principle or any excipient listed in the paragraph 6.1 of the Summary of Product Characteristics (RCP) of Neuraceq®;
* Severe chronic kidney disease (estimated glomerular filtra-tion rate <30 mL/min/1.73 m2);
* Performing a PET/CT or scintigraphic exam within 24 hours;
* Impossibility to lay flat for about 60 minutes;
* New York Heart Association (NYHA) class IV;
* Pregnancy or breastfeeding, women with childbearing po-tential and sexually active not employing highly effective contraceptive methods with a low dependency on the user (from the screening to the end of visit 1), which include: i. abstinence, ii. sexual intercourse only with same-sex part-ners, iii. monogamous relationship with a partner with pri-or vasectomy, iv. intrauterine device, v. combined hormo-nal contraception including estrogens and progesteron-like hormones plus the inhibition of ovulation (oral, intravagi-nal or transdermal), vi. hormonal contraception based on progesterone-like compounds plus the inhibition of ovula-tion (oral, injectable, implantable), viii. intrauterine device with hormone release. The highly effective contraceptive measures above are not required for women made sterile by surgical means (for example through tube ligation, hys-terectomy, bilateral salpingectomy, bilateral ovariectomy) or after the menopause, defined as 12 months of spontane-ous amenorrhea without another clinical cause and with el-evated FSH levels in agreement with the expected values for the menopause. For patients with true abstinence or with just same-sex partners, contraception is not required, as far as this is in line with their preferred and habitual lifestyle. Periodical abstinence (for example, estimate of the timing of ovulation or assessment of body temperature) and coitus interruptus are not acceptable contraceptive methods. If a patient stops to be abstinent, she must use the highly effective contraceptive methods above.

The pregnancy status in women potentially fertile will be checked through the measurement of beta human gonado-tropin on the serum and repeated at the end of the study;

* Participation to a study involving the administration of an experimental drug within 30 days from the screening or 5 half-lives of the study drug, whichever the longest;
* Lack of informed consent or impossibility to complete study procedures.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-26 (Actual); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-01-31 (Estimated)

PRIMARY OUTCOMES:
Agreement between two diagnostic approaches to the diagnosis of AL-CA in patients with a monoclonal protein | 24 months

CONTACTS AND LOCATIONS:
Locations (1):
- Fondazione Toscana Gabriele Monasterio, Pisa, Italy

IPD SHARING:
Plan to Share IPD: Undecided